CLINICAL TRIAL: NCT03071770
Title: A Phase 1, Single-Dose, Open-Label Trial to Evaluate the Pharmacokinetics and Safety of AG-120 in Healthy Male Japanese Subjects Relative to Healthy Male Caucasian Subjects
Brief Title: Japanese Bridging Study of Ivosidenib (AG-120) in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Agios Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AG120-C-006
Record Dates: First submitted 2017-03-02; First posted 2017-03-07 (Actual); Last update posted 2018-01-11 (Actual); Status verified 2018-01

CONDITIONS: Healthy
Keywords: Healthy Volunteers; Japanese; Caucasian
MeSH Terms: interventions — ivosidenib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- ivosidenib (AG-120) (Experimental)
  Interventions: Drug: ivosidenib (AG-120)

INTERVENTIONS:
Drug: ivosidenib (AG-120) — A single-dose of ivosidenib (AG-120) administered in healthy Japanese and Caucasian subjects

SUMMARY:
The purpose of this Phase I, single-dose, open-label trial is to evaluate the pharmacokinetics and safety of ivosidenib (AG-120) in healthy, adult male Japanese and Caucasian subjects. The study plans to evaluate 3 cohorts of a single oral dose of ivosidenib (AG-120) in Japanese and Caucasian subjects. Pharmacokinetic sampling will take place serially through-out the duration of subject participation.

ELIGIBILITY:
Inclusion Criteria:

* Applicable to Japanese Subjects Only: Japanese subjects must have been born in Japan, have both parents and grandparents of Japanese origin, and not have lived outside of Japan for more than 5 years.
* Applicable to Caucasian Subjects Only: Non-Japanese subjects must be Caucasian (ie, White) but may be of any ethnicity.
* Healthy male subjects between 18 and 55 years of age (inclusive).
* Provision of voluntary, written informed consent.
* Capable of adhering to trial restrictions and examination schedules, in the opinion of the Investigator.
* Must be able to communicate with the Investigator.
* Must be in good health as determined by the Investigator according to past medical history, physical examination, vital signs, clinical laboratory test results, and ECGs.
* Must have a body mass index (BMI) between 18 and 29 kg/m2 (inclusive), and body weight between 50-120kg.
* Clinical laboratory test results (serum chemistry, hematology, and urinalysis) must be within normal limits or considered by the Investigator to be not clinically significant after confirmation with the Agios Medical Monitor.
* Vital signs (systolic and diastolic blood pressure, pulse rate, and oral body temperature) will be assessed in the supine position after the subject has rested for at least 5 minutes. Subject must be afebrile with vital signs within the following ranges at screening, Day -1 and pre dose: Systolic blood pressure: 90 to 140 mmHg; Diastolic blood pressure: 50 to 90 mmHg; Pulse rate: 40 to 110 bpm
* Must have a normal or clinically acceptable 12-lead ECG no later than Day -1. Subjects must have a pre-dose QT interval corrected for heart rate using Fridericia's formula (QTcF) value or average of 3 values, ≤450 msec. An ECG may be repeated once to determine subject eligibility after confirmation with the Agios Medical Monitor.
* Subjects (with or without vasectomy) must agree to abstain from sexual intercourse or agree to the use of highly effective contraceptive methods (at screening and throughout the course of the trial) and should avoid fathering a child during the course of the trial and for 90 days following the dose of the IMP. Subjects must refrain from sperm donations for the entire duration of the trial and for 90 days following the dose of AG 120.

Exclusion Criteria:

* Any significant medical condition, laboratory abnormality, or psychiatric illness that would prevent the subject from providing informed consent or participating in the trial in the opinion of the Investigator.
* Any condition, including the presence of laboratory abnormalities, which places the subject at an unacceptable risk if he were to participate in the trial.
* Recent history (within 3 years prior to dosing) of any clinically significant neurological, gastrointestinal, renal, hepatic, cardiovascular, psychological, pulmonary, metabolic, endocrine, hematological, or other major disorder.
* Use of any prescribed systemic or topical medication within 30 days or 5 terminal half-lives, whichever is longer, of IMP administration.
* Exposure to an investigational drug within 30 days prior to IMP administration or 5 half lives of that investigational drug, if known (whichever is longer).
* Use of any non-prescribed systemic or topical medication (including vitamin/mineral supplements, and herbal medicines, eg, St. John's Wort) within 7 days of IMP administration.
* Any surgical or medical condition that could affect drug absorption, distribution, metabolism, or excretion (eg, gastrectomy and cholecystectomy)
* Subjects who plan to have any elective or medical procedures during the conduct of the trial (eg, dental procedure).
* History of clinically significant multiple drug allergies (ie, 2 or more).
* Any clinically significant allergic disease.
* History of drug abuse (as defined by the current version of the Diagnostic and Statistical Manual [DSM]) within 2 years prior to IMP administration, or positive drug screen test due to illicit drugs at any time prior to IMP administration during the screening period.
* History of alcohol abuse within 2 years prior to IMP administration, or positive alcohol screen at any time prior to IMP administration during the screening period.
* History of smoking within 3 months prior to IMP administration, or positive urine cotinine screen at any time prior to IMP administration during the screening period.
* Known to have human immunodeficiency virus (HIV), hepatitis, or known to be a carrier of the hepatitis B surface antigen (HBsAg) or hepatitis C antibody (HCV Ab), or have positive results at screening.

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2017-03-31 (Actual); Primary Completion 2017-05-09 (Actual); Study Completion 2017-09-06 (Actual)

PRIMARY OUTCOMES:
AUC | Pharmacokinetic sampling for ivosidenib (AG-120) will be taken for 504 hours (21 days) after single dose
  AG-120 Area Under the Curve
Cmax | Pharmacokinetic sampling for ivosidenib (AG-120) will be taken for 504 hours (21 days) after single dose
  AG-120 Maximum Plasma Concentration

SECONDARY OUTCOMES:
Incidence of Adverse Events | 28 days after single-dose ivosidenib (AG-120)
  Assessment of adverse events

CONTACTS AND LOCATIONS:
Overall Officials: Medical Affairs Agios Pharmaceuticals, Inc, Study Chair — Agios Pharmaceuticals, Inc.
Locations (1):
- West Coast Clinical Trial (WCCT), Cypress, California, United States

IPD SHARING:
Plan to Share IPD: No